CLINICAL TRIAL: NCT03135821
Title: Randomized Placebo Controlled Trial of Traditional Chinese Medicine for Treatment of Irritable Bowel Syndrome
Brief Title: Traditional Chinese Medicine for Treatment of Irritable Bowel Syndrome
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Singapore College of Traditional Chinese Medicine (Unknown); Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SGH-TCM-GASTR-TCMIBS
Record Dates: First submitted 2016-10-31; First posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Placebo vs Traditional Chinese Medication (TCM) Drug A,B,C,D
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 10% active Placebo (Placebo Comparator): Placebo will constitute granules with 10% active core ingredients as below:
  White Peony Root 10g Processed Liquorice 3g Immature Bitter Orange 8g White Atractylodes Rhizome 15g
  - 2 packets of sachets once before breakfast and once before dinner.
  Interventions: Diagnostic Test: TCM
- Traditional Chinese Medication (TCM) Drug A,B,C,D (Active Comparator): Traditional Chinese Medication (TCM) Drug A,B,C,D.
  TCM Drug A:
  White Peony Root 10g Processed Liquorice 3g Immature Bitter Orange 8g White Atractylodes Rhizome15g
  TCM Drug B:
  White Peony Root 10g Processed Liquorice 3g Immature Bitter Orange 8g White Atractylodes Rhizome 15g Liver stagnation with heaty transformation: add Scutellaria Root 5g、Prunella Spike 5g
  TCM Drug C:
  White Peony Root 10g Processed Liquorice 3g Immature Bitter Orange 8g White Atractylodes Rhizome 15g Prominent abdominal pain: White Peony Root to increase to 15g add Bupleurum Root 5g
  TCM Drug D:
  White Peony Root 10g Processed Liquorice 3g Immature Bitter Orange 8g White Atractylodes Rhizome 15g Hard stools: add Peach Kernel 5g、Areca Seed 5g
  Interventions: Diagnostic Test: TCM

INTERVENTIONS:
Diagnostic Test: TCM

SUMMARY:
Irritable bowel syndrome (IBS) is a prevalent condition that adversely affects patient's quality of life and represents a large health care burden globally. Currently, there is no satisfactory treatment for IBS and Chinese Herbal medicine (CHM) has been suggested to be potentially useful. However, the efficacy of CHM in the treatment of IBS is unclear and its mechanism of action is unknown. To date, attempts to characterize CHM efficacy universally suffer from poor scientific method or they do not faithfully replicate authentic CHM best practice. The overall goal of this proposal is hence to address these deficiencies by combining the best of CHM with western medicine.The investigators propose a 10-week randomized, double-blind, placebo-controlled study on 104 patients that form the intersect between western medicine and CHM. The participants would fulfill ROME III criteria for IBS-Constipation predominant subtype, which is also the TCM (Traditional Chinese Medicine) syndrome of Liver Qi stagnation. The investigators will test a core herbal formula specific for treatment of Liver Qi stagnation against placebo that consist of only 10% active ingredients but which is indistinguishable by taste from active treatment. Efficacy will be assessed by comparing symptoms reported at baseline (2-week run-in period) to end of treatment (8 weeks) and an optional follow up period (12 weeks). The primary end point will be improvement in IBS-Symptom Severity Score. Mechanism of action will be explored by measuring changes to the stool microbiome and GI transit times. If successful, this trial would provide one of the first evidence- and mechanism-based approach to translate CHM into mainstream IBS management.

DETAILED DESCRIPTION:
This will be a 10 week randomized, double blind, parallel group, single center study on patients who fulfil ROME III criteria for IBS-Constipation predominant subtype (IBS-C) and TCM syndrome of Liver Qi stagnation.The study will consist of a two week baseline run-in period without medication, an 8 week randomized double blind treatment period with either placebo or CHM (twice daily), followed by an optional further 12 week withdrawal period with no medication.

Patients who fulfill ROME III criteria for IBS-C will be assessed by a designated qualified traditional Chinese physician. Patients who fulfill TCM syndrome diagnosis of Liver Qi stagnation will be eligible participate in the study.

Each patient's TCM syndrome differentiation and modifications as well as corresponding prescription will be assessed by a second TCM physician to evaluate for reproducibility of TCM diagnosis.

The TCM physician will prescribe the appropriate treatment formula based on TCM principles (see intervention section):

Placebo will constitute granules with 10% active core ingredients. This choice of placebo has been validated in a thesis which showed that the decoction compounded this way was indistinguishable by an intelligent sensory machine in taste, smell and appearance compared to the active treatment formula while not possessing any significant therapeutic effect in animal models

The herbal formulas will be provided in the form of an identical packet of granules for each patient. The patient will be dissolved the granules in water before taking. The patient needs to take one packet of the assigned formulation per time and 2 times a day for the next 8 weeks. The formula will be fixed throughout the 8 week treatment period.

At screening, patients will provide blood for routine testing (FBC,UECr,LFT,PT,APTT and ECG). Patients' medications will be screened and patients instructed to discontinue any medications drugs which may alter GI motility or microbiota (eg: opioids, prokinetics and antibiotics). except bisacodyl).Patients are allowed to take bisacodyl when abdominal pain or discomfort ≥7 on an 11-point numeric rating scale. Data from patient's symptoms during the 2 run-in weeks will be used as the baseline. The subjects will visit the study site at the start and end of the baseline screening period (days 0 and 14), week 4 of during the treatment, end of treatment (week 8), and at the end on the 12 week follow up period. During all these visits, they will be evaluated by the primary investigators and our TCM collaborators. At the end of 4 weeks of treatment, patient's TCM syndrome will be reassessed by the TCM physician to evaluate for mid treatment changes. The diagnosis will performed by a second TCM physician to check for reproducibility. In addition, the patients will be contacted by phone or email weekly to monitor treatment compliance and symptoms. Where necessary, the use of rescue medication bisacodyl 5 mg tablets will be allowed and the quantity of usage will be recorded weekly.

In order to assess mechanisms associated with the patients symptom changes, two approaches will be adopted. First, whole and regional GI transit times will be assessed using the wireless motility capsule. Second, CHM and/or placebo associated changes to the resident bacterial populations, or microbiome, in GI will be assessed by deep sequencing the hypervariable regions of the 16s gene. Patients will be advised not to change their usual diet and exercise level during the trial as this has been shown to alter gut microbiome and motility. The patients' baseline and end of treatment diet will be assessed on weeks 2 and 10 respectively by means of a 3 days food diary (2 week day and 1 weekend day) with verbal and written instructions explaining that they should add to their diary every time they eat or drink, describing the food as accurately as possible and giving estimates of amounts. The completed food records would be evaluated and analysed by the dietician. The patients' exercise levels will be assessed with a validated questionnaire, International physical activity questionnaire(IPAQ) Efficacy assessments and end points

The following symptoms will be recorded: worst abdominal pain (an 11-point numeric rating scale), abdominal discomfort (an 11-point numeric rating scale), abdominal cramping (an 11-point numeric rating scale), abdominal fullness (an 11-point numeric rating scale), abdominal bloating (an 11-point numeric rating scale), IBS Symptom severity score (IBS-SSS), Quality of life questionnaire EQ-5D, Hospital anxiety depression scale, 15 item Somatic Symptom Severity Scale, the number of BMs, quantity of rescue medication used (bisacodyl 5 mg tablets), TCM IBS symptom score Economic Costs of Functional Gastrointestinal Disorders, IPAQ_English_self-admin, IBSMode Questionnaire, Patient's Diary, Food Diary and .TCM Liver Qi Stagnation.

Each BM was assessed for: sensation of complete bowel emptying (yes/no), stool consistency (7-point Bristol Stool Chart), severity of straining (5-point ordinal scale).

ELIGIBILITY:
Inclusion Criteria:

* Ethnic group: Chinese only
* Presence of FGID as determined by managing physician and fulfil ROME III criteria for IBS-C
* To be eligible for randomization, patients will need to report during the baseline period:

  o IBS-symptom severity score (SSS) of ≥150
* Physical examination without clinically relevant abnormalities
* Completed a relevant colonic imaging (e.g. colonoscopy, barium enema, or other colonic imaging) within 60 months before enrolment that shows absence of structural abnormality which could account for the patient's symptom as determined by the managing physician

  o Patients below the age of 45 without colonic imaging must have stable IBS-C symptoms for at least 5 years (without evidence of rectal bleeding, weight loss, recent changes in bowel habits, family history of colorectal cancer or anaemia)
* Completed blood test

  * Haemoglobin within range of 11-17g/dL (for females), and 13-19g/dL (for males) Abnormal haemoglobin which is accounted for by a non-GI-related condition (e.g. thalassemia), as determined by managing physician, is allowed
  * Blood tests taken 3 months or longer before enrolment are considered invalid
* Completed 12-Lead ECG

  * No clinically relevant abnormalities in 12-lead ECG performed for this study and in laboratory findings
  * 12-Lead ECG taken 3 months or longer before enrolment are considered invalid
* Oral contraceptives are allowed provided that they have not been changed in the previous 6 months before the start of the run-in period
* The patient has the ability to provide informed consent
* Patient is willing to be compliant with study procedures including, and will be contactable by phone for weekly IBS treatment and symptoms
* Mentally competent, able to give written informed consent prior to any study-related procedure and compliant to undergo all visits and procedures scheduled in the study.

Exclusion Criteria:

* BMI <16 or >35 A history of surgery to remove a segment of the gastrointestinal tract or bariatric surgery for obesity at any time; appendectomy/cholecystectomy within 2 months or other abdominal surgeries within 6 months before entry into the trial; history of diverticulitis or any chronic condition that could be associated with abdominal pain or discomfort and could confound the assessments in this trial; or a history of laxative abuse. Investigations for exclusion of structural abnormality will be performed as per regional guideline (19).
* Failure to discontinue medication prior to study, specifically:

  * antibiotics and probiotic consumption within the last 1 month
  * CHM medications within the last 2 weeks
* All medications except bisacodyl (rescue medication) which may alter GI motility will also have to be stopped during the 2 weeks run-in period.

  o Patients are allowed to take rescue medication if in need, when abdominal pain or distension ≥70 on irritable bowel syndrome severity scoring system
* Pregnancy or breastfeeding
* Hypersensitivity to the drug excipients.
* Patient is not able to understand or collaborate throughout the study.
* Not currently or in the preceding 4 weeks enrolled in a clinical study with another investigational drug.
* Patient has any condition that, in the opinion of the Investigator that would compromise the well-being of the patient or the requirements of the study.
* Presence of ischaemic heart disease, diabetes mellitus, thyroid dysfunction or renal impairment (as determined by study investigators) or previous surgery or anatomical anomalies which may alter GI motility (as assessed by investigators)
* Failure to maintain usual diet, lifestyle and exercise regimen throughout the study.
* Patients with major psychiatric or neurological disorders

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in IBS-Symptom Severity Score at 8 weeks | 8 weeks
  Improvement in IBS-Symptom Severity Score

CONTACTS AND LOCATIONS:
Overall Officials: Yu Tien Wang, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Drossman DA, Dumitrascu DL. Rome III: New standard for functional gastrointestinal disorders. J Gastrointestin Liver Dis. 2006 Sep;15(3):237-41. PMID 17013448
- [Result] Li Q, Yang GY, Liu JP. Syndrome differentiation in chinese herbal medicine for irritable bowel syndrome: a literature review of randomized trials. Evid Based Complement Alternat Med. 2013;2013:232147. doi: 10.1155/2013/232147. Epub 2013 Mar 11. PMID 23554827
- [Result] Gwee KA, Bak YT, Ghoshal UC, Gonlachanvit S, Lee OY, Fock KM, Chua AS, Lu CL, Goh KL, Kositchaiwat C, Makharia G, Park HJ, Chang FY, Fukudo S, Choi MG, Bhatia S, Ke M, Hou X, Hongo M; Asian Neurogastroenterology and Motility Association. Asian consensus on irritable bowel syndrome. J Gastroenterol Hepatol. 2010 Jul;25(7):1189-205. doi: 10.1111/j.1440-1746.2010.06353.x. PMID 20594245
- [Result] Saad RJ, Hasler WL. A technical review and clinical assessment of the wireless motility capsule. Gastroenterol Hepatol (N Y). 2011 Dec;7(12):795-804. PMID 22347818
- [Result] Cardol M, de Haan RJ, de Jong BA, van den Bos GA, de Groot IJ. Psychometric properties of the Impact on Participation and Autonomy Questionnaire. Arch Phys Med Rehabil. 2001 Feb;82(2):210-6. doi: 10.1053/apmr.2001.18218. PMID 11239312
- [Result] Francis CY, Morris J, Whorwell PJ. The irritable bowel severity scoring system: a simple method of monitoring irritable bowel syndrome and its progress. Aliment Pharmacol Ther. 1997 Apr;11(2):395-402. doi: 10.1046/j.1365-2036.1997.142318000.x. PMID 9146781
- [Result] Rabin R, de Charro F. EQ-5D: a measure of health status from the EuroQol Group. Ann Med. 2001 Jul;33(5):337-43. doi: 10.3109/07853890109002087. PMID 11491192
- [Result] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Result] Kroenke K, Spitzer RL, Williams JB. The PHQ-15: validity of a new measure for evaluating the severity of somatic symptoms. Psychosom Med. 2002 Mar-Apr;64(2):258-66. doi: 10.1097/00006842-200203000-00008. PMID 11914441
- [Result] Sisson G, Ayis S, Sherwood RA, Bjarnason I. Randomised clinical trial: A liquid multi-strain probiotic vs. placebo in the irritable bowel syndrome--a 12 week double-blind study. Aliment Pharmacol Ther. 2014 Jul;40(1):51-62. doi: 10.1111/apt.12787. Epub 2014 May 11. PMID 24815298